CLINICAL TRIAL: NCT06638359
Title: Effects of an Acute Bout of Moderate-Intensity Aerobic Exercise And High-Intensity Intermittent Exercise On Sleep During Night Shifts In Medical Shift Workers With Sleep Impairment: A Single-Blind Crossover Randomized Controlled Trial
Brief Title: Effects of Moderate Exercise And Interval Exercise On Sleep Quality
Acronym: EX&sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chih-Hui Chiu, Professor, National Taiwan Sport University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 113-6; 113-3 (Other: NTUS)
Record Dates: First submitted 2024-09-18; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Exercise Addiction; Control Condition
Keywords: Heart rate variability; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: The effects of a single bout of moderate- aerobic continuous exercise (MACE) and high-intensity intermittent exercise (HIIE) on sleep during continuous night shifts in medical shift workers with mild sleep impairment.
Who Masked: Investigator
Masking Description: control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Experimental): moderate intensity or interval exercise
  Interventions: Behavioral: moderate exercise; Behavioral: interval exercise; Behavioral: Control (placebo) group
- control (Sham Comparator): without exercise
  Interventions: Behavioral: moderate exercise; Behavioral: interval exercise; Behavioral: Control (placebo) group

INTERVENTIONS:
Behavioral: moderate exercise — moderate exercise for 47 minutes
Behavioral: interval exercise — interval exercise for 28 minutes
Behavioral: Control (placebo) group — without exercise

SUMMARY:
This study aimed to explore the effects of a single bout of moderate- aerobic continuous exercise (MACE) and high-intensity intermittent exercise (HIIE) on sleep during continuous night shifts in medical shift workers with mild sleep impairment.

DETAILED DESCRIPTION:
Medical staff with sleep disturbances due to their night-shift work were randomized to either a treadmill walking session for 47 minutes with moderate intensity (the heart rate reaches 70~75% of the maximum heart rate), treadmill running section for 28 minutes with intermittent high-intensity (the heart rate reaches 90~95% of the maximum heart rate for 4 minutes and 50~70% for 3 minutes), or a quiet-rest control, 14 hours before undertaking a continuous night shift. Sleep quality was assessed by ActiGraph with subjective questionnaire for 1 night and 3 nights after exercise. Tests were performed (t-tests or χ2 tests) to test for differences between any two of the three intervention trials.

ELIGIBILITY:
Inclusion Criteria:

* medical staff who have worked at least three consecutive night shifts
* reporting sleep disturbed during the night shift
* not taking sleep/psychotropic medications
* no clinical diagnosis of sleep apnea or other sleep disorder
* not exercising regularly

Exclusion Criteria:

* not medical staff
* without night shift
* taking sleep/psychotropic medications
* exercising regularly

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
total sleep time | Day 1
  total sleep time on Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sport research center, Principal Investigator — National Taiwan University of Sport
Locations (1):
- National Taiwan University of Sport, Taichung, North, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

DOCUMENTS (1):
  • Study Protocol (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT06638359/Prot_000.pdf